CLINICAL TRIAL: NCT00769626
Title: Standardizing Management of Patients With Low Back Pain in Primary Care and Physical Therapy: A Randomized Clinical Trial
Brief Title: Standardizing Management of Patients With Low Back Pain in Primary Care and Physical Therapy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Unable to recruit patients
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Julie M. Fritz, Clinical Outcomes Research Scientist, Intermountain Healthcare
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DES-529-2008
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Last update posted 2011-07-18 (Estimated); Status verified 2008-10

CONDITIONS: Back Pain; Low Back Pain
Keywords: Low Back Pain; Clinical Practice Guidelines; Spinal Manipulation; Physical Therapy Techniques
MeSH Terms: conditions — Back Pain; Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early Treatment (Experimental)
  Interventions: Other: Early Treatment
- Usual Care (Active Comparator)
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Usual Care — Patients in the usual care group will receive advice and education to remain active and anticipate a favorable prognosis. Patients will also receive medication from the primary care provider consistent with current evidence-based guidelines(acetaminophen or non-steroidal anti-inflammatories). Consistent with current practice guidelines, patients will be instructed to return to the primary care provider if they are not satisfied with their progress after 4 weeks.
  Arms: Usual Care
Other: Early Treatment — Patients in the early treatment group will receive the usual care intervention (advice and education, and medication consistent with current evidence-based guidelines). Patients will also be referred to physical therapy for 4 sessions over a 3-week period. A standardized protocol will be used in physical therapy including spinal manipulation and trunk strengthening exercises. Patients will be instructed to return to the primary care provider if they are not satisfied with their progress after completion of the 4 sessions.
  Arms: Early Treatment

SUMMARY:
The purpose of this study is to compare the clinical outcomes and costs associated with two different management strategies for patients with acute low back pain who consult their primary care physician. The investigators hypothesize that management using a brief, standardized physical therapy intervention will result in better outcomes than management based on current practice guideline recommendations of watchful waiting for the first 4 weeks following consultation.

DETAILED DESCRIPTION:
The Institute of Medicine recognizes low back pain (LBP) as a top 15 priority condition, calling for health care organizations to develop new, evidence-based management strategies. Most patients with acute LBP are managed in primary care. Primary care management is characterized by high variability in decision-making, including referral to specialties such as physical therapy. In the face of this variability it is not surprising that the outcomes of management for patients with acute LBP are also inconsistent, with a considerable proportion going on to persistent or recurrent symptoms. Costs associated with patients who fail to recover quickly or completely can be substantial.

Many patients with acute LBP are referred from primary care to physical therapy. Physical therapy management of patients with acute LBP is also highly variable in terms of the interventions used and the outcomes achieved. More effective and standardized management for patients with acute LBP could impact progression of the condition before the concerns associated with chronic pain become evident, and are therefore central to reducing costs and improving outcomes.

Numerous practice guidelines have been developed to attempt to reduce variability and improve outcomes for patients with acute LBP managed in primary care. Current guidelines provide little direction for determining the optimal type of patient and timing for referral to physical therapy, other than a broad recommendation to delay referral for at least a few weeks. Within physical therapy there is an absence of validated decision-support tools to reduce inappropriate variation in care and improve outcomes. The Investigators have developed and validated a clinical decision rule identifying a subgroup of patients with LBP likely to experience rapid and sustained improvement with a brief, standardized physical therapy intervention delivered early in the course of care, suggesting it may be more cost-effective to manage this subgroup with early referral to physical therapy. The impact of integrating this rule into routine clinical care has not been assessed.

We will conduct a randomized clinical trial examining outcomes and costs associated with integrating the decision rule into primary care management of patients with LBP. Patients with LBP who fit the decision rule criteria will be randomized into one of two groups; one managed with usual care based on current practice guidelines; the other managed based on the decision rule with early, standardized physical therapy. Patients will be followed for 6 months. Outcomes will include measures of disability, pain, satisfaction, and costs.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of pain and/or numbness between the 12th rib and buttocks with or without symptoms into one or both legs, which, in the opinion of the primary care provider, originate from the lumbar region.
* Age 18 - 60 years
* Oswestry disability score > 20%
* Both of the clinical decision rule criteria: Duration of current symptoms < 16 days, and patient report of no symptoms (pain, numbness, etc.) distal to the knee since onset.

Exclusion Criteria:

* Prior surgery to the lumbosacral spine
* Current pregnancy
* Neurogenic LBP defined as the presence of either: a positive straight leg raise test (symptom reproduction at <450) or reflex, sensory, or strength consistent with lumbar nerve root compression
* Judgment of the primary care provider of "red flags" of a potentially serious condition including cauda equina syndrome, major or rapidly progressing neurological deficit, fracture, cancer, or infection

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2008-09; Primary Completion 2009-09 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Questionnaire Patient Global Rating of Improvement | 6 months

SECONDARY OUTCOMES:
Numeric Pain Rating Scale Fear-Avoidance Beliefs Questionnaire Patient Satisfaction Questionnaire European Quality of Life (EuroQOL) Direct medical costs | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Julie M Fritz, PhD,PT,ATC, Principal Investigator — Intermountain Healthcare, The University of Utah; Gerard P Brennan, PhD, PT, Study Director — Intermountain Health Care, Inc.
Locations (3):
- United States (3):
  - Intermountain Healthcare, South Jordan Health Center, South Jordan, Utah
  - Intermountain Healthcare Taylorsville Health Center, Taylorsville, Utah
  - Intermountain Healthcare West Jordan Health Center, West Jordan, Utah